CLINICAL TRIAL: NCT04867863
Title: SCREENING OF CELIAC DISEASE IN SCHOLAR CHILDREN IN ITALY
Status: Completed | Type: Observational
Sponsor: Università Politecnica delle Marche (Other)
Collaborators: FONDAZIONE CARIVERONA (Unknown); Azienda ULSS di Verona e Provincia (Other)
Responsible Party: Principal Investigator, Carlo Catassi, M.D., PROFESSOR OF PEDIATRICS AND HEAD OF THE DEPARTMENT OF PEDIATRICS, UNIVERSITA POLITECNICA DELLE MARCHE, Università Politecnica delle Marche
Other Study IDs: 121CELIA14
Record Dates: First submitted 2021-04-27; First posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Celiac Disease; Dental Caries
Keywords: celiac disease; children; caries; HLA DQ2; HLA DQ8; screening
MeSH Terms: conditions — Celiac Disease; Dental Caries

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The main aim of the study is to currently define the prevalence of celiac disease (CD) in children aged 5-10 years in 2 Italian cities (Ancona and Verona). The screening protocol is based on a 1st line genetic test (searche of HLA DQ2/DQ8 genotypes) followed by a serological diagnosis (IgA TTG and IgG DGP).

DETAILED DESCRIPTION:
All scholar children aged 5-10 years living in the cities of Ancona and Verona will be invited to partecipate. Children enrolled will be investigated as follows:

1. HLA DQ2/DQ8 genotyping (by a rapid test)
2. In children genetically predisposed to CD serological investigations will be performed (both IgA TTG and IgG DGP antibodies)
3. The overall population will be evaluated for the prevalence and severity of dental caries (by using the DMFT/dmft index)

ELIGIBILITY:
Inclusion Criteria: age 5-10 -

Exclusion Criteria: celiac disease, on a gluten free diet

-

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 5-10 years
Sampling Method: Probability Sample
Enrollment: 4570 (Actual)
Dates: Start 2015-05; Primary Completion 2016-02 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
prevalence of celiac serology in children aged 5-10 | 2 years

SECONDARY OUTCOMES:
prevalence of dental caries in children genetically predisposed to CD in comparison with children not predisposed | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatrics Universita' Politecnica Delle Marche, Ancona, Italy